CLINICAL TRIAL: NCT05484999
Title: The Maternal Well-Being Study: A Feasibility and Acceptability Trial of Postpartum Support Interventions
Brief Title: The Maternal Well-Being Study
Acronym: MWB
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: A22-4290
Record Dates: First submitted 2022-06-16; First posted 2022-08-02 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Postpartum Depression; Postpartum Anxiety; Weight Retention, Postpartum; Nutritional and Metabolic Diseases
Keywords: nutrition; postpartum; perinatal mood disorders; medically-tailored meals
MeSH Terms: conditions — Depression, Postpartum; Gestational Weight Gain; Nutritional and Metabolic Diseases | interventions — Meals

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dual interventions (Experimental): Receive both interventions: MamaMeals and MamaMatters Interventions
  Interventions: Other: Meals; Other: Meals + Social Support
- Meals intervention only (Active Comparator): MamaMeals
  Interventions: Other: Meals
- Control (Sham Comparator): Wait-list control (received MamaMeals between 16-20 weeks postpartum) (after primary data collection time point)
  Interventions: Other: Control

INTERVENTIONS:
Other: Meals — 12 weeks of medically tailored meals
  Other Names: MamaMeals
  Arms: Dual interventions; Meals intervention only
Other: Meals + Social Support — 12 weeks of medically tailored meals and12 weeks of social media based support
  Other Names: MamaMeals + MamaMatters
  Arms: Dual interventions
Other: Control — Waitlist Control Group (no intervention for first 4 months and then receive MamaMeals between 16-20 weeks postpartum)
  Arms: Control

SUMMARY:
This project aims to understand the local feasibility and acceptability of MamaMeals (a home-delivered nutritious, postpartum meal delivery program) and MamaMatters (a moderated social media-based peer support group) among peripartum women who are eligible for federal supplemental nutrition assistance programs such as The Special Supplemental Nutrition Program for Women, Infants and Children (WIC) or Supplemental Nutrition Assistance Program (SNAP). The investigators will conduct a prospective randomized controlled trial (RCT) of these two interventions among postpartum individuals. Analyses will be performed to determine the relative risk of postpartum depressive or anxiety symptoms (primary outcome) and overall well-being and maternal/infant health (secondary/exploratory outcomes) between groups. Findings from this pilot intervention study will inform a future, large RCT exploring the effectiveness of MamaMeals and/or MamaMatters on reducing postpartum mental health symptoms and cardiovascular morbidity among individuals with food insecurity during and after pregnancy.

DETAILED DESCRIPTION:
1. To assess the local feasibility and acceptability of MamaMeals (home-delivered, nutritious meals) during the 4th trimester for mothers with peripartum food insecurity.
2. To explore perceptions about receiving a medically-tailored meal delivery intervention during the 4th trimester (MamaMeals) among a diverse sample of peripartum individuals with food insecurity (FI).
3. To assess through a randomized trial the potential efficacy of the MamaMeals (nutritious, home-delivered meals) and MamaMatters (ehealth postpartum support) interventions on peripartum mood disorders (primary outcome), postpartum cardiometabolic risk* (exploratory outcome), maternal wellbeing (exploratory outcome), and infant health (exploratory outcome) during the first 12 months following delivery. Hypothesis: Individuals who receive the MamaMeals + MamaMatters interventions will have lower Edinburgh Postpartum Depression Scale (EPDS) scores throughout the first 12 weeks postpartum compared to groups receiving only one intervention or the control group.

ELIGIBILITY:
Inclusion Criteria:

* screen positive for food insecurity or qualify for any of the following governmental assistance programs Medicaid, WIC, SNAP, TANF,
* speak English,
* are between 20-40 completed weeks of pregnancy,
* are ages 18 years or older.

Exclusion Criteria:

* type 1 diabetes
* dietary contraindications (e.g., severe food allergy, or inflammatory bowel disease, celiac disease, chronic renal disease, bariatric surgery, short bowel syndrome)
* an active eating disorder (self-reported)
* hospitalization in the past 12 months for a mental health concern
* a history of postpartum psychosis
* Individuals with a history of being banned from any social media site will also be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2022-05-16 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
% of meals delivered to and consumed by subjects | 12 weeks
  Feasibility of meal delivery social media support delivery
perception of the nutritious home delivered meal program | 12 weeks
  subject engagement with interventions and perception of interventions

SECONDARY OUTCOMES:
% of Edinburgh postnatal depression scale score >15 at 12 weeks postpartum | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Tech University Health Sciences Center, Amarillo, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided